CLINICAL TRIAL: NCT01569685
Title: The Treatment of Traumatised Refugees With Sertraline Versus Venlafaxine in Combination With Psychotherapy - a Randomised Clinical Study
Brief Title: The Treatment of Traumatised Refugees With Sertraline Versus Venlafaxine in Combination With Psychotherapy
Acronym: PTF3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charlotte Sonne (Other)
Collaborators: Psychiatric Center Ballerup (Other)
Responsible Party: Sponsor-Investigator, Charlotte Sonne, Clinical assistent, MD, Psychiatric Center Ballerup
Organization: Psychiatric Center Ballerup (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTF3
Record Dates: First submitted 2012-03-28; First posted 2012-04-03 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Post Traumatic Stress Disorder; Depression
Keywords: PTSD; Traumatic Stress; Depressions; Refugees
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Venlafaxine Hydrochloride; Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Venlafaxine (Active Comparator): 6 months treament vith Venlafaxine (if patient has troubles sleeping in combination with Mianserine) in recommended dose in combination with Cognitive Behavioral Therapy
  Interventions: Drug: Venlafaxine
- Sertraline (Active Comparator): 6 months treament vith Sertraline (if patient has troubles sleeping in combination with Mianserine) in recommended dose in combination with Cognitive Behavioral Therapy
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Venlafaxine — Tablets, once a day, max 375 mg day (maximal recommended dose)
  Other Names: Efexor
  Arms: Venlafaxine
Drug: Sertraline — Tablets, once a day, maximum 200 mg/day (maximum required dose)
  Arms: Sertraline

SUMMARY:
Background: The treatment of traumatised refugees is one of the areas within the field of psychiatry with the weakest evidence for the different types of treatment. This is a problem for both patients and doctors as well as for society.

The treatment of choice today for Post Traumatic Stress disorder (PTSD) is antidepressants from the subgroup of Selektive Serotonin Reuptake Inhibitors (SSRI), among these the drug Sertraline. The evidence for the use of these drugs as treatment for chronically complex PTSD in traumatised refugees is however very limited and a large part of the group is estimated to be insufficiently treated with this type of medicine. Venlafaxine is an antidepressant from the subgroup of dual action product which means that is works on several pathways in the brain. Among others it influences the area in the brain that is responsible for the enhanced anxiety and hyperarousal experienced by traumatised refugees and which is found to be enlarged among patients suffering from PTSD.

All together there is not sufficient evidence to conclude which type of medical and psychological treatment that is most efficient when it comes to the treatment of traumatised refugees. Also there is a lack of studies which examines social functioning and the relation between psychosocial resources and outcome from treatment. Furthermore there is a lack of knowledge of predictors of treatment outcome for the individual patients. This study seeks to produce some of this evidence.

Method: This study is expected to include approximately 150 patients randomised into two different groups. The patients are treated with Setraline or Venlafaxine depending on the group the randomised to. Patients in both groups are getting the same version of manual based Cognitive Behavioural Therapy that is specially adapted to this group of patients. The treatment period is 6-7 month. The trial endpoints are PTSD-and depression symptoms and social functioning all measured on internationally validated ratings scales.

Furthermore the study will examine the relation between expected outcome of treatment from a range of predictors and the actual treatment results for the individual patient.

Results: Altogether this study will bring forward new standards for clinical evaluation and treatment of traumatised refugees and the results are expected to be used in reference programmes/clinical guidelines.

DETAILED DESCRIPTION:
Please see the summary above

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to treatment in Psychiatric Clinic for refugees, Psychiatric Center Ballerup between April 2012 to May 2013
* Adults (18 years or older)
* Refugees or reunified with a refugee spouse
* Symptoms of PTSD defined by ICD-10 research criterias.
* Previosly traumatized
* Motivated for treatment
* Informed consent

Exclusion Criteria:

* Psychotic disorder (ICD-10 diagnosis F2x og F30.1-F309)
* Active substance abuse (ICD-10 F1x.24-F1x.26).
* In need of acute admission to psychiatric hospital)
* No informed consent
* Pregnant women, breastfeeding women or women who wish to become pregnant within the project period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Harvard Trauma Questionnaire (HTQ) | Change from baseline after aprox. 6 months treatment
  Self administered Rating Scale

SECONDARY OUTCOMES:
Hopkins Symptom Check List (HSCL-25) | Change from baseline after aprox. 6 months treatment
Social Adjustment Scale Self Report (SAS-SR) short version | Change from baseline after aprox. 6 months treatment
Hamilton Depresssion Scale (17 items) | Change from baseline after aprox. 6 months treatment
Hamilton Anxiety Scale (14 items) | Change from baseline after aprox. 6 months treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte K Sonne, MD, Principal Investigator — Psychiatric Center Ballerup
Locations (1):
- Competence Center for Transcultural Psychiatry, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Sonne C, Carlsson J, Bech P, Elklit A, Mortensen EL. Treatment of trauma-affected refugees with venlafaxine versus sertraline combined with psychotherapy - a randomised study. BMC Psychiatry. 2016 Nov 8;16(1):383. doi: 10.1186/s12888-016-1081-5. PMID 27825327
- [Derived] Sonne C, Carlsson J, Elklit A, Mortensen EL, Ekstrom M. Treatment of traumatized refugees with sertraline versus venlafaxine in combination with psychotherapy - study protocol for a randomized clinical trial. Trials. 2013 May 11;14:137. doi: 10.1186/1745-6215-14-137. PMID 23663588